CLINICAL TRIAL: NCT01534182
Title: A 6-month, Randomized, Active Comparator, Open-label, Multi-Center Study to Evaluate Patient Outcomes, Safety and Tolerability of (Fingolimod) 0.5 mg/Day in Patients With Relapsing Remitting Multiple Sclerosis Who Are Candidates for Multiple Sclerosis (MS) Therapy Change From Previous Disease Modifying Therapy (DMT)
Brief Title: Evaluation of Patient Reported Outcomes in RRMS Patients Candidates for MS Therapy Change and Transitioned to Fingolimod 0.5 mg (EPOC)
Acronym: EPOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DRU01
Record Dates: First submitted 2012-02-08; First posted 2012-02-16 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis (RRMS); Fingolimod; Disease Modifying Therapy (DMT); TSQM-9
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride; Interferon beta-1a; Glatiramer Acetate

ARMS (2):
- Fingolimod (Experimental): Participants received 0.5 mg orally once a day.
  Interventions: Drug: Fingolimod
- Standard Disease Modifying Therapy (DMT) (Active Comparator): Participants received interferon beta-1a (IFN), 44 mcg subcutaneously 3 times a week or glatiramer acetate (GA), 20 mg subcutaneously once a day.
  Interventions: Drug: Interferon beta - 1a (IFN); Drug: Glatiramer acetate (GA)

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg orally once a day
  Other Names: Gilenya
  Arms: Fingolimod
Drug: Interferon beta - 1a (IFN) — 44 mcg subcutaneously three times a week
  Other Names: Rebif
  Arms: Standard Disease Modifying Therapy (DMT)
Drug: Glatiramer acetate (GA) — 20 mg subcutaneously once a day
  Other Names: Copaxone
  Arms: Standard Disease Modifying Therapy (DMT)

SUMMARY:
A 6-month, Randomized, Active Comparator, Open-label, Multi-Center Study to Evaluate Patient Outcomes, Safety and Tolerability of (fingolimod) 0.5 mg/day in Patients with Relapsing Remitting Multiple Sclerosis who are candidates for MS therapy change from Previous Disease Modifying Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Patients must be diagnosed with relapsing remitting MS (RRMS) as defined by 2005 revised McDonald criteria (McDonald et al 2001, Polman et al 2005) (Appendix 2).
* Patients who explicitly agree to be assigned to a treatment group that may receive or DMT after having been informed about their respective benefits and possible adverse events by the investigator.
* Male or female patients aged 18-70 years.
* An Expanded Disability Status Scale (EDSS) score of 0-6 inclusive.
* Must have received continuous treatment with a single approved and indicated MS DMT for a minimum of 6 months prior to the screening visit. Patients must continue with this MS DMT until the randomization visit.
* Naïve to treatment with fingolimod.

Exclusion Criteria:

* A manifestation of MS other than those defined in the inclusion criteria.
* A history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome.
* History of malignancy of any organ system.
* Diagnosis of macular edema during Screening Phase.
* Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS or to have positive HIV antibody test.
* Patients who have received any live or live attenuated vaccines (including for varicella-zoster virus or measles) within 2 months prior to baseline.
* Patients who have received total lymphoid irradiation or bone marrow transplantation.
* History of selected immune system treatments and/or medications.
* Any medically unstable condition, as assessed by the investigator.
* Selected cardiovascular, or hepatic conditions
* Selected abnormal laboratory values.
* Patients with any other disease or clinical condition (including neurologic or psychiatric disorders) which may affect patient enrollment into the study and study medication use by the Investigators' opinion.
* Participation in any clinical research study evaluating another not approved in Russia investigational drug or therapy within 6 months prior to baseline.
* History of hypersensitivity to the study drug or to drugs of similar chemical classes.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Russia (24):
  - Novartis Investigative Site, Arkhangelsk, Russia
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Belgorod
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Khanty-Mansiysk
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saransk
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at screening received standard DMT with either interferon beta-1a or glatiramer acetate from day -30 to day -1.
Pre-assignment Details: Eligible participants were then randomized in a 3:1 ratio to fingolimod or a standard DMT. For participants who were randomized to the standard DMT group, those who received IFN during screening were switched to GA at randomization and those who received GA during screening were switched to IFN at randomization.
Period: Overall Study
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Started | 230 | 68
Safety Set | 230 | 64
Full Analysis Set | 229 | 62
Completed | 218 | 58
Not Completed | 12 | 10
Not completed — Administrative problems | 1 | 0
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Adverse Event | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT) | Total
Number analyzed (Participants) | 230 | 68 | 298
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (9.9) | 36.4 (9.3) | 35.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 50 | 212
  Male | 68 | 18 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Treatment Satisfaction
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) contains 14 items assessing the following 4 domains: effectiveness (items 1 - 3), side effects (items 4 - 8), convenience (items 9 - 11) and global satisfaction (items 12 - 14). The primary outcome was measured on the global satisfaction domain. Item 12 scored as 1 (not at all confident) to 5 (extremely confident); item 13 scored as 1 (not at all certain) to 5 (extremely certain); and item 14 scored as 1 (extremely dissatisfied) to 7 (extremely satisfied). Responses to items were summed and transformed: specifically, TSQM v 1.4 domain scale scores were computed by adding the items loading on each domain. The lowest possible score was subtracted from the composite score and divided by the greatest possible score range. This provided a transformed score between 0 and 1 that was then multiplied by 100. The final transformed score ranges from 0 to 100, with higher scores indicating better treatment satisfaction.
Time Frame: Baseline, 6 months
Population: Full Analysis Set (FAS): This set included all randomized participants who had taken at least one dose of study medication and had at least one post-baseline assessment of the TSQM. The last observation carried forward (LOCF) method was applied.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Number analyzed (Participants) | 229 | 62
scores on a scale | 22.69 (28.12) | 13.92 (30.63)

2. Secondary Outcome: Number of Patients Who Experienced Adverse Events, Serious Adverse Events and Death
Description: Participants were monitored for adverse events, serious adverse events and death throughout the study.
Time Frame: 6 months
Population: Safety Set: This set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Number analyzed (Participants) | 230 | 64
Participants
  Adverse events (serious and non-serious) | 73 | 26
  Serious adverse events | 2 | 0
  Deaths | 0 | 0

3. Secondary Outcome: Changes in Patient-reported Effectiveness, Side Effects and Convenience
Description: TSQM v 1.4 domains for effectiveness, side effects and convenience were used to evaluate this outcome. The effectiveness domain for items 1 - 3 was scored as: 1 (extremely dissatisfied) to 7 (extremely satisfied). For the side effects domain, item 4 scored as 0(no) or 1(yes); item 5 scored as 1 (extremely bothersome) to 5 (not at all bothersome); and items 6 - 8 scored as 1 (a great deal) to 5 (not at all). For the convenience domain, items 9 and 10 scored as 1(extremely difficult) to 7 (extremely easy), and item 11 scored as 1 (extremely inconvenient) to 7 (extremely convenient). For each domain, scale scores were computed by adding the items loading on each domain. The lowest possible score was subtracted from the composite score and divided by the greatest possible score range. This provided a transformed score between 0 and 1 that was then multiplied by 100. The final transformed score ranges from 0 to 100, with higher scores indicating better treatment satisfaction.
Time Frame: Baseline, 6 months
Population: FAS: The LOCF method was applied.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Number analyzed (Participants) | 229 | 62
scores on a scale
  Effectiveness | 21.57 (24.01) | 11.56 (20.70)
  Side effects | 26.75 (35.83) | 13.07 (40.19)
  Convenience | 25.38 (20.72) | 10.57 (20.93)

4. Secondary Outcome: Change in Patient-reported Depression
Description: The Beck Depression Inventory (BDI-I) scale was used to measure this outcome. The scale consists of 21 items to assess the intensity of depression in clinical and normal patients. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. Each item was scored from 0 - 3. If more than one score was provided for an item, the maximum score was considered the item score. The total score was calculated as the sum of all individual items and then compared to a key to determine the depression's severity. The standard key ranges were: 0 - 9 indicated minimal depression; 10 - 18 indicated mild depression; 19 - 29 indicated moderate depression and 30 - 63 indicated severe depression. Higher total scores indicate more severe depressive symptoms.
Time Frame: Baseline, 6 months
Population: FAS: The LOCF method was applied.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Number analyzed (Participants) | 229 | 62
scores on a scale | -2.88 (6.80) | -1.86 (8.04)

5. Secondary Outcome: Change in Patient-reported Health-related Quality-of-life Using the Short Form Health Survey v2 Acute (SF-36 v2 Acute)
Description: The SF-36 is a health-related quality of life instrument used in numerous disease states, including MS (Brazier et al 1992). It is a self-administered survey that measures 8 domains of health including: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and general mental health. Two summary scale scores can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each domain was scored by adding the individual items from the domain and transforming the resulting scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Time Frame: Baseline, 6 months
Population: Participants from the full analysis set were considered for this analysis. However, for a given time frame, participants analyzed had both baseline and 6 month asssessment values.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT)
Number analyzed (Participants) | 229 | 62
scores on scale
  Physical functioning (n=225,61) | 3.62 (16.23) | 1.39 (14.23)
  Role limitations due to physical health (n=226,61) | 6.50 (21.99) | 4.30 (27.52)
  Bodily pain (n=225,61) | 5.24 (23.79) | 0.93 (22.95)
  General health (n=226,61) | 4.28 (17.72) | 4.43 (22.57)
  Vitality (n=226,61) | 7.72 (18.61) | 1.95 (21.97)
  Social functioning (n=226,61) | 5.59 (23.36) | 1.64 (23.77)
  Role limit. due to emotional problems (n=224,61) | 7.18 (25.98) | 5.33 (27.00)
  Mental health (n=226,61) | 5.60 (18.55) | 2.79 (22.09)
  Physical component summary (n=222,61) | 1.51 (5.69) | 0.68 (6.57)
  Mental component summary (n=222,61) | 3.16 (9.66) | 1.68 (11.31)

ADVERSE EVENTS:
Groups:
- Standard Disease Modifying Therapy (DMT): Interferon Beta-1a: Participants received interferon beta-1a (IFN), 44 mcg subcutaneously 3 times a week
- Standard Disease Modifying Therapy: Glatiramer Acetate: Patients who received glatiramer acetate (GA), 20 mg subcutaneously once a day.
Arm/Group | Fingolimod | Standard Disease Modifying Therapy (DMT): Interferon Beta-1a | Standard Disease Modifying Therapy: Glatiramer Acetate
Serious Adverse Events (participants affected / at risk) | 2/230 | 0/28 | 0/36
Other Adverse Events (participants affected / at risk) | 39/230 | 13/28 | 10/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=230) | Standard Disease Modifying Therapy (DMT): Interferon Beta-1a (N=28) | Standard Disease Modifying Therapy: Glatiramer Acetate (N=36)
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=230) | Standard Disease Modifying Therapy (DMT): Interferon Beta-1a (N=28) | Standard Disease Modifying Therapy: Glatiramer Acetate (N=36)
Lymphopenia (Blood and lymphatic system disorders) | 27 | 0 | 2
Gamma-Glutamyltransferase increased (Investigations) | 13 | 1 | 0
Alanine aminotransferase increased (Investigations) | 11 | 2 | 0
Influenza like illness (General disorders) | 0 | 10 | 0
Injection site pain (General disorders) | 0 | 1 | 6
Injection site erythema (General disorders) | 0 | 0 | 3
Injection site extravasation (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.